CLINICAL TRIAL: NCT03156426
Title: Prognostic Biomarkers For Acute Kidney Injury In Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC16143
Record Dates: First submitted 2017-02-22; First posted 2017-05-17 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Acute Kidney Injury; Liver Cirrhoses; Biomarkers
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood:
  Haematology: FBC, INR Biochemistry: U&E, LFT Plasma - biomarkers: KIM-1 Urine - proteinuria, fractional excretion of sodium Urinary biomarkers - KIM-1, L-FABP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: Adults with a histological, clinical or radiological diagnosis of cirrhosis who are admitted to RIE over a 4-month period will be approached by a member of their clinical care team for potential participation. Eligible patients may be recruited from accident and emergency, the acute medical unit, hepatology ward, high dependency or intensive care units. Recurrent admissions are common, so only the first admission for each recruited patient will be included. Patients will be monitored to identify acute kidney injury (AKI) during admission.
  Interventions: Other: Event of interest: Acute kidney injury

INTERVENTIONS:
Other: Event of interest: Acute kidney injury — AKI as defined by AKIN staging

SUMMARY:
Acute kidney injury (AKI) is a common and under-diagnosed problem in patients with liver cirrhosis, and is associated with significant illness and preventable death. Blood (serum) creatinine is the current test for kidney function, but it is an insensitive and non-specific marker in cirrhosis. The investigators hypothesise that blood (plasma) levels of kidney injury molecule-1 (KIM-1) will detect AKI earlier and predict the risk of worsening AKI in cirrhosis, thus identifying patients in need of prompt and effective treatment and improving patient outcomes. The investigators will collect blood and urine samples from cirrhosis patients admitted into hospital and study the relationship between plasma KIM-1, other diagnostic 'biomarker' tests that have recently been proposed, and patient outcomes.

DETAILED DESCRIPTION:
In 2015 the International Club of Ascites redefined AKI in cirrhosis as an increase in serum creatinine (sCr) of 26.5 µmol/L as even small increases in sCr are clinically relevant and associated with poorer outcomes. The investigators recently conducted a ward-based study of 105 cirrhotic patients admitted to the Royal Infirmary of Edinburgh (RIE) Liver Unit over a 3-month period and showed that 40% of patients developed AKI, and incidence of AKI increased with severity of cirrhosis. Increased AKI stage was associated with incrementally longer hospital stay, at an extra cost to the NHS of ~£400/day (data.gov.uk), and a greater mortality. Indeed, the mortality rate for cirrhotic patients without AKI was 6%, compared to 18%, 35% and 50% in patients with AKI stage 1, 2 and 3 respectively.

sCr is a suboptimal marker of renal dysfunction in advanced cirrhosis. Despite a normal sCr, patients may already have significant renal dysfunction, thus rendering sCr a late marker of AKI. Moreover, recurrent mild episodes of AKI, where sCr may not exceed normal laboratory limits, can lead to a gradual deterioration in baseline renal function, increased susceptibility to further acute insults and higher mortality. There is an urgent unmet need for a superior, more sensitive biomarker (a renal equivalent of troponin I (TnI)) to better identify cirrhotic patients who are most at risk of developing AKI, to aid earlier recognition of kidney impairment and allow rapid and targeted treatment. This is especially important because pre-transplant renal dysfunction in patients with cirrhosis is associated with increased morbidity and mortality after liver transplantation.

The urinary biomarkers neutrophil gelatinase-associated lipocalin (NGAL), interleukin-18 (IL-18), kidney injury molecule-1 (KIM-1), liver-type fatty acid binding protein (L-FABP) and albumin, are significantly higher in cirrhotic patients with acute tubular necrosis (ATN), compared with pre-renal AKI and hepatorenal syndrome (HRS). Additionally, L-FABP is a marker of renal hypoxia and has been identified as a promising marker for early diagnosis of AKI, and for predicting dialysis requirement and in-hospital mortality. In view of the progressive renal vasoconstriction that occurs as cirrhosis advances, L-FABP may be a potentially relevant marker, although increased hepatic release may render it non-specific in the context of acute liver injury.

Plasma KIM-1 is a biomarker that is specific and sensitive for both acute and chronic kidney injury. KIM-1 is a transmembrane glycoprotein that is upregulated in proximal tubular cells during AKI. Work from our Group showed that early measurement of plasma KIM-1 was a more sensitive predictor of patient outcome than sCr in AKI after paracetamol-induced acute liver injury. Furthermore, in a cohort of patients with type-1 diabetes, normal sCr and normo/microalbuminuria, an elevated plasma KIM-1 level was strongly associated with risk of early progressive renal decline. However, plasma KIM-1 has never been evaluated in patients with chronic liver disease.

HYPOTHESES

1. Plasma KIM-1 will be higher in patients with cirrhosis who go on to develop AKI and serve as an earlier predictive marker when compared with sCr.
2. Plasma KIM-1 will be more effective at early identification of AKI than other candidate AKI biomarkers (fractional excretion of sodium (FeNa), protein to creatinine ratio (PCR), urinary L-FABP and urinary KIM-1).

Protocol

Blood and urine samples will be collected on admission and day 2, to assess initial trends (in a similar way to TnI). Measurements will be repeated on day 7 (or at discharge if <7 days) as a potential indicator of unresolved AKI. Final follow-up samples will be taken 30 days after discharge. Plasma will be prepared from whole blood samples according to an established SOP and stored along with urine specimens (using a linked anonymised format) at -800 d.c. in the RIE Clinical Research Facility (RIE CRF). KIM-1 will be measured by microsphere-based Luminex technology, as previously described for human plasma. Urinary L-FABP will be measured by ELISA. Outcome data up to 30 days will be collected from TRAK and case note reviews.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult subjects over 18 years of age
2. Able to provide written informed consent and able to understand and willing to comply with the requirements of the study
3. Clinical/imaging-diagnosed or biopsy-proven liver cirrhosis of any aetiology
4. Not previously enrolled in this study on a previous admission

Exclusion Criteria:

1) Those patients who do not have capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This exploratory study will test recruitment, sample collection, assess size of change and inform power calculations for a larger Scottish multi-centre study.
  Adults with a histological, clinical or radiological diagnosis of cirrhosis who are admitted to RIE over a 3-month period will be approached by a member of their clinical care team for potential participation. Eligible patients may be recruited from the acute medical unit, hepatology ward, high dependency or intensive care units.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Plasma level of kidney injury molecule-1 (KIM-1) to predict risk of developing AKI - a novel biomarker of early kidney injury | 30 days
  Plasma KIM-1 is a biomarker of kidney damage. We will measure it on admission and analyse the relationship between admission plasma KIM-1 level and risk of developing AKI during hospital stay.

SECONDARY OUTCOMES:
Plasma level of kidney injury molecule-1 (KIM-1) to identify AKI on admission | 30 days
  Plasma KIM-1 is a biomarker of kidney damage. We will measure it on admission and analyse the relationship between plasma KIM-1 level and the presence of AKI on admission.
Plasma level of kidney injury molecule-1 (KIM-1) to identify patients with a greater risk of mortality | 30 days
  Plasma KIM-1 is a biomarker of kidney damage. We will measure it on admission and assess the relationship between plasma KIM-1 level on admission and all-cause mortality rate at day 30
Rate of change in plasma level of kidney injury molecule-1 (KIM-1) between admission and day 2 to predict risk of AKI | 30 days
  We will measure plasma KIM-1 on admission, day 1 and day 2 and assess if there is a relationship between change in plasma KIM-1 level (admission + day 2) and risk of developing AKI.
Fractional excretion of sodium (FeNa): a measurement is taken of urine sodium and creatinine concentration, and compared to serum creatinine and sodium to analyse the degree to which the kidneys are retaining sodium | 30 days
  FeNa has been suggested as a suitable marker of AKI in patients with liver cirrhosis. We will use this as a comparative biomarker to plasma KIM-1 at predicting risk of AKI during hospital stay
Protein-creatinine ratio (PCR): The ratio of protein to creatinine in the urine | 30 days
  PCR is the current gold-standard biomarker for chronic kidney disease and can be helpful in the acute setting. We will compare the performance of PCR with plasma-KIM-1 level on admission at predicting the risk of developing AKI during hospital stay
Urinary liver-fatty acid binding protein (urinary L-FABP) | 30 days
  urinary L-FABP is another novel biomarker which has been suggested as a marker of kidney ischaemia. We will compare the diagnostic performance of urinary L-FABP to plasma- KIM-1 for predicting AKI during admission
Urinary kidney injury molecule-1 (KIM-1) | 30 days.
  Urinary levels of KIM-1 increase during AKI for the same reasons that plasma levels of KIM-1 rise. We will compare whether plasma or urinary KIM-1 is more accurate at predicting AKI during admission

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan A Fallowfield, PhD, Principal Investigator — MRC Centre for Inflammation Research, Queens Medical Research Institute
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual patient data will be available to other researchers